CLINICAL TRIAL: NCT02983656
Title: Analysis on AEFI Surveillance Data for Live Attenuated Varicella Vaccine
Status: Completed | Type: Observational
Sponsor: Zhejiang Provincial Center for Disease Control and Prevention (Other Government)
Collaborators: Changchun Keygen Biological Products Co., Ltd. (Other)
Responsible Party: Principal Investigator, Qian Li, Deputy chief physician, Zhejiang Provincial Center for Disease Control and Prevention
Other Study IDs: ZJCDC20161121
Record Dates: First submitted 2016-12-01; First posted 2016-12-06 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Varicocele
Keywords: Vaccine Safety
MeSH Terms: conditions — Varicocele

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: live attenuated varicella vaccine

SUMMARY:
The purpose of this study is to observe the occurrence of adverse events of live attenuated varicella vaccine.

ELIGIBILITY:
Inclusion Criteria:

* The registered permanent residence or resident place are local (reside more than 3 months);
* Participant preventive inoculation of varicella vaccine in 2014-2015;
* Adverse reactions occurred and should be reported in the AEFI monitoring system.

Exclusion Criteria:

* Subjects with a known allergy to any ingredient of the vaccine, and with any allergy history to any vaccine;
* Subjects with any acute diseases, severe chronic diseases, acute bout of chronic diseases, and catching cold and fever;
* Subjects with uncontrolled seizures and other progressive neurological diseases, with a history of Guillain-Barré syndrome.

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participant preventive inoculation of varicella vaccine in 2014-2015
Sampling Method: Non-Probability Sample
Enrollment: 394 (Actual)
Dates: Start 2016-11; Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
incidence of adverse reactions | 1 year after the first and second doses

CONTACTS AND LOCATIONS:
Overall Officials: Qian Li, Bachelor, Principal Investigator — Zhejiang Provincial Center for Disease Control and Prevention

IPD SHARING:
Plan to Share IPD: No